CLINICAL TRIAL: NCT04449094
Title: Socio-demographic Factors and Emergence of the COVID 19 Epidemic in the City of Nice in 2020
Brief Title: Emergence of the COVID 19 Epidemic in the City of Nice
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20dspcovid01
Record Dates: First submitted 2020-06-25; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive analysis of the appearance of the first cases of COVID 19 diagnosed in the city of Nice. Analysis of the association of socio-demographic factors with the viremia attack rate according to the district of residence.

ELIGIBILITY:
Inclusion Criteria:

* People resident in city of Nice at the COVID diagnosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents in the city of Nice
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Attack rate | 1 month
  Diagnosed cases of COVID 19 divided by the population by district and multiplied by 100,000

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France